CLINICAL TRIAL: NCT03972657
Title: A Phase 1/2 Study of REGN5678 (Anti-PSMAxCD28) With or Without Cemiplimab (Anti-PD-1) in Patients With Metastatic Castration-Resistant Prostate Cancer and Other Tumors Associated With PSMA Expression
Brief Title: A Trial to Find Out if REGN5678 (Nezastomig) is Safe and How Well it Works Alone or in Combination With Cemiplimab for Adult Participants With Metastatic Castration-Resistant Prostate Cancer and Other Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R5678-ONC-1879
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC); Clear Cell Renal Cell Carcinoma (ccRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cemiplimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mCRPC - dose escalation cohort (Experimental): REGN5678 with or without cemiplimab
  Interventions: Drug: REGN5678; Drug: Cemiplimab
- mCRPC - dose expansion cohort (Experimental): REGN5678 with or without cemiplimab
  Interventions: Drug: REGN5678
- ccRCC - dose escalation cohort (Experimental): REGN5678 with or without cemiplimab
  Interventions: Drug: REGN5678; Drug: Cemiplimab
- ccRCC - dose expansion cohort (Experimental): REGN5678 with or without cemiplimab
  Interventions: Drug: REGN5678

INTERVENTIONS:
Drug: REGN5678 — Administered as per the protocol
  Other Names: Nezastomig
Drug: Cemiplimab — Administered as per the protocol
  Other Names: REGN2810; LIBTAYO
  Arms: ccRCC - dose escalation cohort; mCRPC - dose escalation cohort

SUMMARY:
The main purpose of this study is to determine the safety, tolerability (how the body reacts to the drug[s]) and effectiveness (ability to treat the cancer) of REGN5678 (Nezastomig) alone, or in combination with cemiplimab.

The study has 2 parts. The goal of Part 1 (dose escalation) is to determine a safe dose(s) of REGN5678 when it is given alone or in combination with cemiplimab. The goal of Part 2 (dose expansion) is to use the REGN5678 drug dose(s) found in Part 1 to see how well REGN5678 alone or in combination with cemiplimab works to shrink tumors.

This study is looking at several other research questions, including:

1. Side effects that may be experienced by taking REGN5678 alone or in combination with cemiplimab
2. How REGN5678 alone or in combination with cemiplimab works in the body
3. How much REGN5678 and/or cemiplimab are present in the blood
4. To see if REGN5678 alone or in combination with cemiplimab works to reduce the size of the tumor by helping the immune system destroy the tumor

ELIGIBILITY:
Key Inclusion Criteria:

mCRPC cohorts (men):

1. Men with histologically or cytologically confirmed adenocarcinoma of the prostate without pure small cell carcinoma.
2. PSA value at screening ≥4 ng/mL that has progressed within 6 months prior to screening as defined in the protocol.
3. Has received ≥2 lines prior systemic therapy approved in the metastatic and/or castration-resistant setting (in addition to Androgen Deprivation Therapy [ADT]) including at least:

   1. one second-generation anti-androgen therapy (eg, abiraterone, enzalutamide, apalutamide, or darolutamide)
   2. 177Lu-PSMA-617 radiotherapy, or another lutetium-based PSMA targeted radioligand, as described in the protocol

ccRCC cohorts (men and women):

1. Histologically or cytologically confirmed RCC with a clear-cell component.
2. Diagnosis of metastatic ccRCC with at least one measurable lesion via RECIST 1.1 criteria
3. Has progressed on or after ≥1 line prior systemic therapy approved in the metastatic setting. Prior treatment must include an anti-Programmed Death-1 (receptor) [PD-1]/Programmed Death-Ligand 1 (PD-L1) therapy and either ipilimumab and/or a tyrosine kinase inhibitor

Key Exclusion Criteria:

1. Has received treatment with an approved systemic therapy within 3 weeks of dosing or has not yet recovered (ie, grade ≤1 or baseline) from any acute toxicities, as described in the protocol
2. Has received any previous systemic biologic therapy within 5 half-lives of first dose of study therapy, as described in the protocol
3. Has received prior PSMA-targeting therapy with the exception of a PSMA targeting radioligand (eg. 177Lu-PSMA-617) in mCRPC
4. Dose Escalation: Has had prior anti-cancer immunotherapy (other than sipuleucel-T) within 5 half-lives prior to study therapy.
5. Dose Expansion (mCRPC only): Has had prior anti-cancer immunotherapy, as described in the protocol
6. Any condition that requires ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or anti-inflammatory equivalent) within 1 week prior to the first dose of study therapy
7. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, as described in the protocol
8. Encephalitis, meningitis, neurodegenerative disease (with the exception of mild dementia that does not interfere with Activities of Daily Living [ADLs]) or uncontrolled seizures in the year prior to first dose of study therapy
9. Uncontrolled infection with Human Immunodeficiency Virus (HIV), hepatitis B or hepatitis C infection; or diagnosis of immunodeficiency

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) | Through study completion, up to 5 years
  Dose Escalation Phase
Incidence and severity of Adverse Event of Special Interests (AESIs) | Through study completion, up to 5 years
  Dose Escalation Phase
Incidence and severity of Serious Adverse Events (SAEs) | Through study completion, up to 5 years
  Dose Escalation Phase
Number of participants with Grade ≥3 laboratory abnormalities | Through study completion, up to 5 years
  Dose Escalation Phase
Incidence of Dose-Limiting Toxicities (DLTs) | First dose through day 42 of last participant in each dose level
  Dose Escalation Phase
Concentration of REGN5678 in serum over time | Through study completion, up to 5 years
  Dose Escalation Phase
Concentration of REGN5678 in combination with cemiplimab in serum over time | Through study completion, up to 5 years
  Dose Escalation Phase
Composite Response Rate (CRR) of 50% decline of Prostate Specific Antigen (PSA) and/or confirmed radiographic response of complete (CR) or partial response (PR) | Through study completion, up to 5 years
  Dose Expansion Phase - mCRPC cohort
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | Through study completion, up to 5 years
  Dose Expansion Phase - ccRCC cohort

SECONDARY OUTCOMES:
CRR of 50% decline of PSA and/or confirmed radiographic of CR or PR | Through study completion, up to 5 years
  Dose Escalation Phase - mCRPC cohort
ORR per RECIST 1.1 criteria | Through study completion, up to 5 years
  Dose Escalation Phase - ccRCC cohort
Incidence and severity of TEAEs | Through study completion, up to 5 years
  Dose Expansion Phase
Incidence and severity of AESIs | Through study completion, up to 5 years
  Dose Expansion Phase
Incidence and severity of SAEs | Through study completion, up to 5 years
  Dose Expansion Phase
Number of participants with grade ≥3 laboratory abnormalities | Through study completion, up to 5 years
  Dose Expansion Phase
Concentration of REGN5678 in serum over time | Through study completion, up to 5 years
  Dose Expansion Phase
Concentration of REGN5678 in combination with cemiplimab in serum over time | Through study completion, up to 5 years
  Dose Expansion Phase
Percentage of participants with ≥50% decline of PSA | Through study completion, up to 5 years
  Dose Escalation and Dose Expansion Phases - mCRPC cohorts
Percentage of participants with ≥90% decline of PSA | Through study completion, up to 5 years
  Dose Escalation and Dose Expansion Phases- mCRPC cohorts
Presence or absence of antibodies against REGN5678 | Through study completion, up to 5 years
  Dose Escalation and Dose Expansion Phases
Presence or absence of antibodies against cemiplimab | Through study completion, up to 5 years
  Dose Escalation and Dose Expansion Phases

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Management, Study Director — Regeneron Pharmaceuticals
Locations (21):
- United States (21):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - John Wayne Cancer Institute (JWCI), Santa Monica, California
  - Sarah Cannon Research Institute (SCRI), Denver, Colorado
  - Yale University Hospital, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center - McKinley Drive, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University - The Trustees of Columbia University in the City of New York, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of Rochester Medical Center (URMC) - Wilmot Cancer Institute (WCI) (James P. Wilmot Cancer Center) - Rochester, Rochester, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health & Science University (3485 S. Bond), Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
  - MD Anderson Cancer Center, Houston, Texas
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/